CLINICAL TRIAL: NCT02749227
Title: Pilot Study of Pasireotide LAR Treatment of Silent Corticotrophin Pituitary Tumors and Effects on Plasma Levels of POMC
Brief Title: Pasireotide LAR Therapy of Silent Corticotroph Pituitary Tumors
Acronym: PASSILCORT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine at the Columbia University Medical Center, Dept of Medicine Endocrinology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ6255; CSOM230GUS44T (Other: Novartis)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-03

CONDITIONS: Pituitary Tumor; ACTH-producing Pituitary Tumour
Keywords: Clinically non-functioning pituitary adenomas (CNFAs); silent corticotroph adenomas
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pasireotide LAR Therapy (Experimental): Subjects will receive Pasireotide LAR monthly. Safety labs and Pituitary MRI will be performed.
  Interventions: Drug: Pasireotide LAR

INTERVENTIONS:
Drug: Pasireotide LAR — Pasireotide LAR (SIGNIFOR® LAR) is a somatostatin analog indicated for the treatment of patients with acromegaly who have had an inadequate response to surgery and/or for whom surgery is not an option. It is a long acting release injectable suspension for intramuscular use.
  The starting dose is Pasireotide LAR 40 mg/month intramuscular (IM), this will be increased to 60 mg/month at 6 months if a fall in POMC levels and/or tumor shrinkage are not attained.
  Other Names: Signifor LAR

SUMMARY:
This is a phase II, open-label, 12-month pilot study in 10 patients with silent corticotroph pituitary tumors testing the hypotheses that Pasireotide long-acting release (LAR) treatment of patients with silent corticotroph pituitary tumors and elevated plasma Proopiomelanocortin (POMC) levels will reduce plasma POMC levels and this will be associated with a reduction in pituitary tumor size. Pasireotide LAR 40 mg will be administered monthly. Baseline and monthly visits on therapy will monitor plasma levels of POMC, other pituitary function, safety labs, glucose tolerance, physical examination, and visual fields. Pituitary magnetic resonance imaging (MRI) will be done at baseline, 6 months and 12 months of therapy. The eligible patient population will consist of adult patients with known silent corticotroph pituitary tumors and elevated plasma levels of POMC.

DETAILED DESCRIPTION:
Clinically non-functioning pituitary adenomas (CNFAs), the subtype of pituitary adenomas that does not appear to secrete biologically active hormone nor to have a characteristic clinical phenotype, are the most common type of pituitary macroadenoma at diagnosis. There is currently no option for medical therapy of CNFA, in general, or specifically of silent corticotroph tumors. Silent corticotroph tumors can range from being completely asymptomatic to becoming large and causing significant hypothalamic/pituitary dysfunction and visual symptoms, and most data support that this type of tumor has a more aggressive phenotype. Current therapy consists primarily of surgical removal of the tumor and for recurrent or residual tumors, repeated surgery and/or radiotherapy. In very aggressive tumors, chemotherapy has been tried with some success. Therefore, a need exists for a medical therapeutic option for the treatment of this tumor type. This project assesses this clinical need.

ELIGIBILITY:
Inclusion criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Adults (males and females) with a diagnosis of a clinically nonfunctioning pituitary tumor of the silent corticotroph tumor type (i.e., positive adrenocorticotropin (ACTH) staining on immunohistochemical staining of the pituitary tumor obtained at surgery)
2. Plasma POMC level > upper limit of normal
3. Prior pituitary tumor surgery with residual or recurrent pituitary tumor visible on MRI scan that is ≥ 5 mm from the optic chiasm.
4. Surgical resection of the pituitary adenoma must have occurred two or more months prior to enrollment
5. If patients have undergone pituitary radiotherapy they must have completed their course of radiotherapy at least 2 months prior to study screening
6. No prior somatostatin analog therapy
7. No concurrent use of dopamine agonist therapy
8. No active malignancy
9. Stable pituitary hormone supplements (x 2 months) prior to baseline visit
10. Sign and date an informed consent document indicating that the subject has been informed of and agrees to all pertinent aspects of the trial

Exclusion criteria:

Subjects must not meet any of the following exclusion criteria to be eligible for enrollment into the study:

1. Patients with Cushing's disease (biochemical evidence of hypercortisolism)
2. Patients with compression of the optic chiasm causing any visual field defect that requires surgical intervention
3. Diabetic patients with poor glycemic control as evidenced by HbA1c >8%
4. Patients who are hypothyroid or adrenally insufficient and not on adequate replacement therapy
5. Patients with symptomatic cholelithiasis and acute or chronic pancreatitis
6. Patients with risk factors for torsade de pointes, i.e., patients with a baseline QTcF (Fridericia's Correction Formula value) >450 ms in males, and >460 ms in females
7. Hypokalaemia, hypomagnesaemia, uncontrolled hypothyroidism, family history of long QT syndrome or concomitant medications with known risk of Torsades de pointes (TdP). Drugs with possible risk of TdP should be avoided whenever feasible
8. Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, history of acute myocardial infarction (MI) less than one year prior to study entry or clinically significant impairment in cardiovascular function
9. Concomitant disease(s) that could prolong the QT interval such as autonomic neuropathy (caused by diabetes or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
10. Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with alanine aminotransferase (ALT)/aspartate aminotransferase (AST) > 2.0 X upper limit of normal (ULN), serum bilirubin >2.0 X ULN
11. Presence of Hepatitis B surface antigen (HbsAg) or Hepatitis C antibody test (anti-HCV)
12. Patients with serum creatinine >2.0 X ULN
13. Patients with white blood cell (WBC) count <3 X 109/L; Hb 90% < lower limit of normal (LLN); platelet (PLT) count <100 X 109/L
14. Patients with the presence of active or suspected acute or chronic uncontrolled infection
15. Patients who have undergone major surgery/surgical therapy for any cause within 4 weeks prior screening
16. Patients with abnormal coagulation (PT and/or activated partial thromboplastin time (APTT) elevated by 30% above normal limits) or patients receiving anticoagulants that affect PT (prothrombin time) or APTT (activated partial thromboplastin time)
17. History of syncope or family history of idiopathic sudden death
18. History of immunocompromise, including a positive HIV test result (ELISA and Western blot)
19. Sexually active males unless they use a condom during intercourse while taking drug and for 3 months following last dose of pasireotide and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
20. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
21. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and 3 months following last dose of pasireotide. Highly effective contraception methods include:

    * Total abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject
    * Combination of any two of the following (a+b or a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

         * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
         * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Freda, MD, Principal Investigator — Columbia University
Locations (1):
- Neuroendocrine Unit and Pituitary Center, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pasireotide LAR Therapy: Subjects will receive Pasireotide LAR monthly. Safety labs and Pituitary MRI will be performed.
  Pasireotide LAR: Pasireotide LAR (SIGNIFOR® LAR) is a somatostatin analog indicated for the treatment of patients with acromegaly who have had an inadequate response to surgery and/or for whom surgery is not an option. It is a long acting release injectable suspension for intramuscular use.
  The starting dose is Pasireotide LAR 40 mg/month intramuscular (IM), this will be increased to 60 mg/month at 6 months if a fall in POMC levels and/or tumor shrinkage are not attained.
Period: Overall Study
Arm/Group | Pasireotide LAR Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pasireotide LAR Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Proopiomelanocortin (POMC) Levels
Description: This is to measure the effect of Pasireotide LAR (long-acting release) treatment.
Time Frame: Baseline, 12 months
Population: The study was terminated due to poor enrollment. The data was not collected or analyzed.
Arm/Group | Pasireotide LAR Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Pituitary Tumor Volume
Description: This is to measure the effect of Pasireotide LAR (long-acting release) treatment.
Time Frame: Baseline, 12 months
Population: The study was terminated due to poor enrollment. The data was not collected or analyzed.
Arm/Group | Pasireotide LAR Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Pasireotide LAR Therapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The study was terminated due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT02749227/Prot_SAP_000.pdf